CLINICAL TRIAL: NCT01127971
Title: Patient Registry: A Study of the Use of Accelerated Partial Breast Irradiation to Evaluate Local Tumor Control, Cosmetic Outcome and Toxicities
Brief Title: Patient Registry: Partial Breast Irradiation
Acronym: PBI Registry
Status: Terminated | Type: Observational
Why Stopped: administrative reasons (no impact/concern of subject rights, welfare, safety)
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: L-04-147E
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2014-10

CONDITIONS: Breast Cancer
Keywords: patients; receiving; irradiation; device; External Beam
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — No biospecimens collected
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an Aurora Health Care system registry of patients receiving accelerated partial breast irradiation and external beam.

ELIGIBILITY:
Inclusion Criteria:

* Aurora patients who decide to undergo PBI treatment in the next 5-years or who have had PBI Treatment in the last ten-years. All such patients are female.

Exclusion Criteria:

* Patients not seen in an Aurora facility

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aurora Health Care system patients receiving accelerated partial breast irradiation
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2010-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The collection and analysis of sufficient data to determine 5 and 10-year local recurrence rates is collection and analysis of sufficient data to determine 5 and 10-year local recurrence rates | 5 and 10-year local recurrence rates
  The primary endpoint of this registry trial is collection and analysis of sufficient data to determine 5 and 10-year local recurrence rates for each PBI type used and for the overall Aurora population. The following endpoints will also be reported and analyzed:
  * Disease Free Survival
  * Regional Recurrence
  * Distant Metastasis
  * Combined Recurrence

SECONDARY OUTCOMES:
collection and analysis of data to evaluate and compare cosmetic outcome | 5 and 10-year
  The secondary endpoint is the collection and analysis of data to evaluate and compare cosmetic outcome (per Harvard Score) and toxicities/complications for each PBI type (per Common Terminology Criteria for Adverse Events (referred to as CTC or CTCAE))

CONTACTS AND LOCATIONS:
Overall Officials: David Rohde, MD, Principal Investigator — Aurora BayCare Medical Center
Locations (1):
- Aurora BayCare Medical Center, Green Bay, Wisconsin, United States